CLINICAL TRIAL: NCT03772639
Title: Shared Decision Making and Patient Engagement Program During AECOPD Hospitalization
Brief Title: Shared Decision Making in Hospitalized AECOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0082UG
Record Dates: First submitted 2018-12-05; First posted 2018-12-11 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group received a standard medical and pharmacological care in a daily format and shared decision making (SDM). The general framework of SDM was developed focusing on self-management goals which include education that addresses continuous use of medication, behavioral change, breathing training, learning to interpret changes in the disease and its consequences, and use of medical and community resources.
  Interventions: Other: Shared decision making
- Control Group (No Intervention): The control group received standard care and pharmacological care including systemic steroids, antibiotics, inhaled bronchodilators, and oxygen therapy.

INTERVENTIONS:
Other: Shared decision making — Decision-making processes focused on the knowledge of the disease for set up adjusted care management about their necessities and engaging in recommended health behaviors
  Arms: Experimental group

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a leading cause of morbidity and mortality worldwide. Patients require good communication with the physician to improve control illness. Shared decision making is a promising opportunity for chronic disease management due to the relative cost, medicine optimization and decreases hospital admissions/re-admissions

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the leading one on hospital care cost, physician services, and prescription drugs. Additionally to the disease progression with the reduction in lung function, COPD patients experiment a progressive decline in functional capacity and health-related quality of life (HRQoL) with a significant burden in terms of disability. Shared Decision Making is defined as an approach where clinicians and patients share the available information to making clinical decisions, and where patients are counseled. SDM is a way to empower patients when decisions are made about treatment as a determinant factor in patient-centered care. Decision aids have been proven effective in improving disease knowledge, decision making, and self-care.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were COPD patients hospitalized due to acute exacerbation

Exclusion Criteria:

* Exclusion criteria were the inability to provide informed consent, the presence of psychiatric or cognitive disorders, progressive neurological disorders, organ failure, cancer, or inability to cooperate. Patients who had experienced another exacerbation of COPD in the previous month were also excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | Participants will be followed for the duration of hospital stay, an expected average of 9 days and after discharge 3 months follow up
  European Quality of Life questionnaire consists of the EQ-5D visual analog scale and the EQ-5D index. The visual analog scale has a rating scale of 0-100 (0 worst possible health, and 100 best possible health). The questionnaire has 5 domains: mobility, self-care, usual activity, pain, and anxiety-depression. For each item, the subject selects one of 3 descriptive health states (from good to poor).

SECONDARY OUTCOMES:
COPD Knowledge | Participants will be followed for the duration of hospital stay, an expected average of 9 days and after discharge 3 months follow up
  Chronic Obstructive Pulmonary Disease Questionnaire (COPD-Q). COPD knowledge was evaluated using the Chronic Obstructive Pulmonary Disease Knowledge Questionnaire (COPD-Q; Maples, Franks, Ray, Stevens, & Wallace, 2010). The COPD-Q is a valid, readable, and reliable 13-item (each one score 0 to 3) self-administered true/false questionnaire assessing COPD knowledge in patients with low health literacy skills. A higher punctuation indicates better results.
Adherence of inhalers | Participants will be followed for the duration of hospital stay, an expected average of 9 days and after discharge 3 months follow up
  The Test of Adherence to Inhalers (TAI) was used to assess the level of adherence to inhalers in asthma and COPD patients. The test has two subscores, first to identify non-adherent patients and to measure the non-adherence level, second was designed to guide clinically the treatment non-compliance patients. Low adherence is considered when scores are less than 45 points in the 10-items subscore.
Functional capacity | Participants will be followed for the duration of hospital stay, an expected average of 9 days and after discharge 3 months follow up
  Functional independence was assessed using the Functional Independence Mease Scale (FIM). This scale has 18 items that are grouped into 2 dimensions, 13 motor items, and 5 cognitive items. The total score range between 18 points (total dependence) to 126 points (Independence completes).
Physical activity | Participants will be followed for the duration of hospital stay, an expected average of 9 days and after discharge 3 months follow up
  The International Physical Activity Questionnaire (IPAQ) short form measures walking, moderate- and vigorous intensity, and total PA and daily time spent sitting on weekdays. PA was reported in MET·minutes/week and days per week and was scored using standardized IPAQ scoring protocols to yield total metabolic equivalent minutes (MET·minutes/week) of PA per week. Sitting time was reported as the amount of time in hours and/or minutes participants spent sitting on a weekday during the past seven days.
Nutritional status | Participants will be followed for the duration of hospital stay, an expected average of 9 days and after discharge 3 months follow up
  Nutritional status was assessed with Mini Nutritional Assessment (MNA). The MNA has a screening- and assessment part. The screening part consists of questions about food intake, weight loss, mobility, stress, neuropsychological problems and weight and height will be combined to report BMI in kg/m^2. When the MNA punctuation is ≥ 24 nutritional status can be considered good.
Functional capacity associated with breathlessness | Participants will be followed for the duration of hospital stay, an expected average of 9 days and after discharge 3 months follow up
  Functional capacity associated with breathlessness was assessed with London Chest Activity of Daily Living Scale (LCADL): The LCADL is a 15-item scale divided into 4 domains: self-care (4 items), domestic (6 items), physical (2 items), and leisure (3 items). The use of 0 representing 'I wouldn't do any way' and 5 representing that patients require help.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cross AJ, Thomas D, Liang J, Abramson MJ, George J, Zairina E. Educational interventions for health professionals managing chronic obstructive pulmonary disease in primary care. Cochrane Database Syst Rev. 2022 May 6;5(5):CD012652. doi: 10.1002/14651858.CD012652.pub2. PMID 35514131